CLINICAL TRIAL: NCT05439993
Title: A Phase 1b/2 Study of Tepotinib in Combination With Paclitaxel in Patients With MET Amplified or MET Exon 14 Alterated Advanced Gastric and Gastroesophageal Junction Carcinoma
Brief Title: Tepotinib Plus Paclitaxel in MET Amplified or MET Exon 14 Alterated Gastric and GEJ Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Zang, Dae Young, Professor, Hallym University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tepotinib in GC
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tepotinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tepotinib plus paclitaxel arm (Experimental)
  Interventions: Drug: Tepotinib plus paclitaxel

INTERVENTIONS:
Drug: Tepotinib plus paclitaxel — Paclitaxel 80mg/m2 on D1, 8, 15 tepotinib 250mg or 500mg daily on D1-28 Q 4weeks

SUMMARY:
Purpose of this study is to define the maximal tolerated dose (MTD) and recommended phase 2 dose (RP2D) of paclitaxel and tepotinib combination therapy in patients with advanced tumors and to evaluate the efficacy of paclitaxel and tepotinib combination treatment as second-line therapy in patients with advanced gastric and gastroesophageal junction carcinomas (AGC/GEJCs) with MET amplification or MET exon 14 alterations. This study is devided into Phase 1b and Phase 2 study.

ELIGIBILITY:
Inclusion Criteria:

1. Have the willingness to sign a written informed consent document prior to any study specific precedures
2. Age ≥ 19 years of male and female
3. At each phase of the trial, subjects who meet the following requirements in the appropriate phase will be enrolled.

   A. Phase 1b: Subjects with a histologically confirmed metastatic solid tumor that have progressed after treatment with approved therapies or for which there is no standard effective therapy available.

   B. Phase 2b: Subjects with histologically confirmed locally advanced or metastatic gastric and gastroesophageal carcinoma that have progressed after treatment with first-line fluoropyrimidine-based chemotherapy, with MET amplified (copy number gain ≥3) or MET exon 14 skipping mutation in the archival or fresh tumor tissue specimen identified in study customized targeted DNA deep sequencing (NGS by gastric cancer panel). If the subject received adjuvant chemotherapy after curative gastric resection and lymph node dissection, adjuvant chemotherapy is considered to be the first-line palliative chemotherapy if the disease recurred during adjuvant chemotherapy or within 6 months after the completion of adjuvant chemotherapy.
4. Patients must have measurable disease based on RECIST 1.1 (Phase 2 part only) Measurable disease will not be required for enrollment in the phase1b part. Patients with evaluable lesion only (without measurable lesion) can be enrolled in the phase 1b part.
5. ECOG performance status 0-1
6. Patients must have adequate organ and marrow function as defined below:

Exclusion Criteria:

1. Active central nervous system (CNS) lesions (ie, those with radiologically unstable or symptomatic brain lesions). For those who receive radiation or surgical treatment, the subject can be enrolled if the subject is maintained without evidence of CNS disease progression for more than 4 weeks. However, patients with a leptomeningeal metastasis are excluded.
2. Treatment with any of the following:

   * Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
   * Any cytotoxic chemotherapy from a previous treatment regimen within 14 days. If the subject received an investigational drug from another clinical trial, the subejct can be enrolled after 2 weeks of last administration and more than 5 x half-life of the investigational drug. If monoclonal antibody therapy was given, the subject can be enrolled after four weeks after the last does.
   * Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment. If acute symptoms of radiation have fully resolved, the extent and timing of radiotherapy for eligibility can be discussed between the local investigator and principal investigator.
   * Any previous exposure to a c-MET inhibitor
3. History of allogeneic bone marrow transplantation or organ transplantation
4. History of another primary cancer (excluding gastric cancer):
5. Clinically significant cardiovascular disease including but not limited to:

   * Acute coronary syndome within the 6 months prior to the initiation of study drug (including myocardial infarction or unstable angina, Coronary Artery Bypass Graft surgery, percuatneous coronary intervention and stenting)
   * Current heart failure or past history of heart failure
   * Left ventricle ejection fraction (LVEF) < 50%; if there is no past history of heart failure, screening with echocardiography to confirm EF is not required.
   * Current or past history of clinically significant cardiac arrhythmia (eg, complete left bundle branch block, third degree heart block)
   * Any risk factors that prolong QTc or increase the probability of arrhythmia, including medication (eg: heart failure, hypokalemia, congenital long QT syndrome, history of Torsades de Pointes)
6. Persistent uncontrolled hypertension as defined by: systolic >180 mmHg or diastolic >100 mmHg despite medical treatment
7. Seropositivity of HIV or known active hepatitis B and/or active hepatitis C infection. Hepatitis B carriers may be enrolled if prophylactic use of an antiviral agent with minimal interaction with CYP3A4 is administered to inhibit HBV activation (eg. Entecavir, adefovir)
8. Impairment of gastrointestinal function or gastrointestinal disorders (eg. untreated ulcerative disorders; uncontrolled nausea, vomiting, or diarrhea; absorption disorder syndrome; small bowel resection; ileostomy). Patients with ileostomcy will not allowed to be enrolled, but patients with colostomy can be enrolled to this study.
9. As judged by the Investigator, all other symptoms and associated disease for which the investigator determined that participation in this study is contraindicated (e.g. Infection/inflammation; severe liver dysfunction; bilateral diffuse interstitial lung disease; uncontrolled renal disease; unstable heart and lung disease; hemorrhagic disease; intestinal obstruction; unable to swallow oral pills; social and psychological problems, etc)
10. Pregnant or lactating women. Pregnancy is defined as the state from conception confirmed by HCG clinical laboratory test to termination of pregnancy.
11. Medical, psychiatric, cognitive, or other conditions that may interfere with the ability of the subject to understand the subject information, provide the informed consent, follow the protocol process, or complete the clinical trial
12. Hypersensitivity to paclitaxel

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate (PFSR) at 4 months | PFSR at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, Dr, Principal Investigator — Hally University Medical Center
Locations (1):
- Hallym University Medical Center, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez Garcia D, Grau Mirete B, Rodriguez Paya P, Ferrandez-Arias A, Borregon-Rivilla M, Lazaro-Sanchez AD, Benitez-Fuentes JD. Adding Docetaxel to Tepotinib to Overcome Oligoprogression in MET Exon 14 Skipping-Mutated NSCLC When Local Therapy Is Unfeasible: A Case Report. Case Rep Oncol Med. 2025 Aug 19;2025:4483379. doi: 10.1155/crom/4483379. eCollection 2025. PMID 40880848